CLINICAL TRIAL: NCT05346406
Title: Comparing Peripherally Inserted Central Catheters to Long Peripheral Catheters for Non-central Vascular Access Indications - a Clinical Effectiveness Pilot Trial in Pediatrics
Brief Title: Comparing Peripherally Inserted Central Catheters to Long Peripheral Catheters in Pediatrics
Acronym: ComPLET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Alina Burek, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCW2022
Record Dates: First submitted 2022-04-01; First posted 2022-04-26 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Vascular Access Device Complications
Keywords: peripherally inserted central catheters, long peripheral catheters
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Peripherally Inserted Central Catheter, Randomized (PICC R) (Active Comparator)
  Interventions: Device: Peripherally Inserted Central Catheter
- Midline Catheter, Randomized (MC R) (Experimental): Also known as long peripheral catheter (LPC)
  Interventions: Device: Midline Catheter
- Peripherally Inserted Central Catheter, Non-randomized (PICC NR) (No Intervention): Observational only arm
- Midline Catheter, Non-Randomized (MC NR) (No Intervention): Observational only arm

INTERVENTIONS:
Device: Midline Catheter — Bard Powerglide 8 cm midline catheter
  Other Names: Long peripheral catheter
  Arms: Midline Catheter, Randomized (MC R)
Device: Peripherally Inserted Central Catheter — Bard 3fr, 4fr or 6fr; Cook 4fr; or Medcomp 1.9fr and 2.6fr
  Arms: Peripherally Inserted Central Catheter, Randomized (PICC R)

SUMMARY:
Peripherally Inserted Central Catheters (PICCs) are frequently used in hospitalized children who require prolonged vascular access; however, concerns regarding their inappropriate use and contribution to serious complications such as central line associated blood stream infection (CLABSI) and venous thromboembolism (VTE) have triggered exploration of safer alternatives. Long Peripheral Catheters (LPCs) have been recently adopted by some institutions due to fewer complications as compared to PICCs. The investigators hypothesize that LPCs could be safer alternatives to PICCs for medium-term vascular access (5-14 days) in the appropriate cohort of hospitalized pediatric patients. The primary objective of the proposed clinical effectiveness pilot trial is to test the feasibility of a full-scale effectiveness trial comparing PICCs to LPCs in hospitalized pediatric patients. The investigators aim to identify a population in which LPCs are safe and effective alternatives to PICCs for medium-term, non-central vascular access; data that will inform the design of a full-scale effectiveness study. The investigators plan to engage patients and families as advisors in vascular access device selection by understanding their experience with vascular access device placement and maintenance. Over time, use of LPCs should result in decreased inappropriate PICC utilization with a concomitant decrease in serious complications such as CLABSI and VTE.

DETAILED DESCRIPTION:
Hospitalized children frequently require a vascular access device (VAD) for delivery of life saving interventions such as intravenous fluids and antibiotics. Peripherally Inserted Central Catheters (PICCs) are central VADs frequently used in hospitalized children for prolonged vascular access, or to administer solutions not compatible with peripheral infusion. However, PICC related complications such as venous thromboembolism (VTE) and central line associated blood stream infections (CLABSI) have triggered exploration of safer alternatives. Long Peripheral Catheters (LPCs) are peripheral VADs recently adopted for medium-term vascular access (5-14 days) and peripherally compatible infusate, due to potential for fewer complications compared to PICCs. However, there is a scarcity of literature on the effective and safe use of LPCs in pediatrics. To reduce the use of PICCs when central venous access is not required (i.e., infusate is peripherally compatible), feasible alternatives for vascular access need to be identified and tested. Until clinicians and other stakeholders are given effective alternatives for durable vascular access and evidence-based tools for VAD selection, central VAD related complications will remain a critical concern, placing children at risk for harm and increasing healthcare costs.

The overall objective of this application is to test the feasibility of a full-scale effectiveness trial comparing PICCs to LPCs and identify a population in which a LPC would be a safe and effective alternative to a PICC. In a prior study, our group showed that as many as 139 PICCs over a one-year period were placed at our local institution in children that (1) did not require central venous access for administration of peripherally incompatible infusate, (2) had the VAD in for < 14 days, and (3) did not discharge home with the VAD, but because of PICC placement for vascular access these children were at risk for CLABSI and VTE. The pediatric population satisfying the above conditions is the target of our pilot trial. A LPC program was introduced at our local institution in 2019 with initiation in the intensive care units and plans to expand the program to the whole hospital by the fall of 2021. In our initial group of 20 successfully placed LPCs, there were no severe complications (VTE and CLABSI).

The aims of this pilot, randomized controlled trial are:

Aim 1: To assess the feasibility of a full-scale effectiveness trial comparing PICCs to LPCs in hospitalized pediatric patients in need of non-central, medium-term vascular access (5-14 days anticipated need).

Hypothesis: Feasibility of a full-scale effectiveness trial will be established by demonstrating that > 70% of eligible patients agree to enrollment and randomization, > 80% of randomized patients receive the assigned intervention, > 80% of providers involved find the study acceptable, and < 5% of data are missing.

Aim 2: To identify a population in which a LPC is a safe and effective alternative to a PICC for vascular access in hospitalized pediatric patients age > 2 years, in need of non-central, medium-term access.

Hypothesis: LPCs are non-inferior to PICCs for delivery of peripherally compatible infusate needed for 5-14 days in hospitalized pediatric patients. The investigators plan to determine the time-to-removal of the VAD, both secondary to completion of therapy and secondary to complications. Safety will be assessed by measuring complication rate (e.g., VTE, CLABSI, occlusion, dislodgement, phlebitis).

Aim 3: To engage patients and families as advisors in vascular access device selection.

The investigators will describe the patient and family experience with device placement and maintenance as well as perceived patient and parent insertion-related and sedation-related distress. Mixed methods (quantitative and qualitative analysis) will be used for this aim.

The results of this study will guide the design of a full-scale effectiveness clinical trial comparing PICCs and LPCs in pediatric patients that require medium-term, non-central venous access. The investigators will identify patient characteristics and clinical situations in which LPCs are safe and effective alternatives to PICCs, allowing us to take the next step to reduce PICC use and the associated complications. The family and patient experience with VADs will add essential information that will guide device selection and future research on patient-centered outcomes. Our work will add to ongoing efforts to improve health care quality and safety in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* patients age 2 to 17 years admitted to Children's Wisconsin and requesting placement of a PICC for:

  1. anticipated length of intravenous treatment of 5-14 days AND
  2. peripherally compatible infusate AND
  3. VAD not needed at discharge

Exclusion Criteria:

* non-English-speaking family
* active bacteremia or VTE at site where device would be placed
* urgent need of vascular access (within 4 hours)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Burek, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paterson RS, Chopra V, Brown E, Kleidon TM, Cooke M, Rickard CM, Bernstein SJ, Ullman AJ. Selection and Insertion of Vascular Access Devices in Pediatrics: A Systematic Review. Pediatrics. 2020 Jun;145(Suppl 3):S243-S268. doi: 10.1542/peds.2019-3474H. PMID 32482738
- [Background] Ullman AJ, Marsh N, Mihala G, Cooke M, Rickard CM. Complications of Central Venous Access Devices: A Systematic Review. Pediatrics. 2015 Nov;136(5):e1331-44. doi: 10.1542/peds.2015-1507. Epub 2015 Oct 12. PMID 26459655
- [Background] Ullman AJ, Bernstein SJ, Brown E, Aiyagari R, Doellman D, Faustino EVS, Gore B, Jacobs JP, Jaffray J, Kleidon T, Mahajan PV, McBride CA, Morton K, Pitts S, Prentice E, Rivard DC, Shaughnessy E, Stranz M, Wolf J, Cooper DS, Cooke M, Rickard CM, Chopra V. The Michigan Appropriateness Guide for Intravenous Catheters in Pediatrics: miniMAGIC. Pediatrics. 2020 Jun;145(Suppl 3):S269-S284. doi: 10.1542/peds.2019-3474I. PMID 32482739
- [Background] Gibson C, Connolly BL, Moineddin R, Mahant S, Filipescu D, Amaral JG. Peripherally inserted central catheters: use at a tertiary care pediatric center. J Vasc Interv Radiol. 2013 Sep;24(9):1323-31. doi: 10.1016/j.jvir.2013.04.010. Epub 2013 Jul 19. PMID 23876551
- [Background] Burek AG, Parker J, Bentzien R, Talbert L, Havas M, Hanson SJ. The Development of a Long Peripheral Catheter Program at a Large Pediatric Academic Center: A Pilot Study. Hosp Pediatr. 2020 Oct;10(10):897-901. doi: 10.1542/hpeds.2020-0181. PMID 32998934
- [Background] Noonan PJ, Hanson SJ, Simpson PM, Dasgupta M, Petersen TL. Comparison of Complication Rates of Central Venous Catheters Versus Peripherally Inserted Central Venous Catheters in Pediatric Patients. Pediatr Crit Care Med. 2018 Dec;19(12):1097-1105. doi: 10.1097/PCC.0000000000001707. PMID 30142121
- [Background] Xu T, Kingsley L, DiNucci S, Messer G, Jeong JH, Morgan B, Shutt K, Yassin MH. Safety and utilization of peripherally inserted central catheters versus midline catheters at a large academic medical center. Am J Infect Control. 2016 Dec 1;44(12):1458-1461. doi: 10.1016/j.ajic.2016.09.010. PMID 27908432
- [Background] Chenoweth KB, Guo JW, Chan B. The Extended Dwell Peripheral Intravenous Catheter Is an Alternative Method of NICU Intravenous Access. Adv Neonatal Care. 2018 Aug;18(4):295-301. doi: 10.1097/ANC.0000000000000515. PMID 29847401
- [Background] Kleidon TM, Schults JA, Wainwright C, Mihala G, Gibson V, Saiyed M, Byrnes J, Cattanach P, Macfarlane F, Graham N, Shevill E, Ullman AJ. Comparison of midline catheters and peripherally inserted central catheters to reduce the need for general anesthesia in children with respiratory disease: A feasibility randomized controlled trial. Paediatr Anaesth. 2021 Sep;31(9):985-995. doi: 10.1111/pan.14229. Epub 2021 Jun 21. PMID 34053159
- [Background] Qian SY, Horn MT, Barnes R, Armstrong D. The use of 8-cm 22G Seldinger catheters for intravenous access in children with cystic fibrosis. J Vasc Access. 2014 Sep-Oct;15(5):415-7. doi: 10.5301/jva.5000274. Epub 2014 Jul 4. PMID 25041922
- [Background] Pacilli M, Bradshaw CJ, Clarke SA. Use of 8-cm 22G-long peripheral cannulas in pediatric patients. J Vasc Access. 2018 Sep;19(5):496-500. doi: 10.1177/1129729818761278. Epub 2018 Mar 12. PMID 29529968
- [Background] Paladini A, Chiaretti A, Sellasie KW, Pittiruti M, Vento G. Ultrasound-guided placement of long peripheral cannulas in children over the age of 10 years admitted to the emergency department: a pilot study. BMJ Paediatr Open. 2018 Mar 28;2(1):e000244. doi: 10.1136/bmjpo-2017-000244. eCollection 2018. PMID 29637197

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We had an enrollment goal of 30 participants per each randomized arm. The RCT eligibility was not met.
Groups:
- Peripherally Inserted Central Catheter, Randomized (PICC R): PICC Randomized arm:
  An uncoated polyurethane PICC with an external clamp was placed in the upper arm, and the available sizes were 3 to 6Fr (Bard, Becton Dickinson). The catheter type and size were selected based on IR standard protocol.
- Midline Catheter, Randomized (MC R): MC Randomized arm:
  An uncoated MC with available sizes of 8 cm, 20 to 22G (Powerglide, Becton Dickinson). The catheter size was selected by an inserter based on patient size. All MCs were placed in the upper arm with the tip of the catheter ending at or below the axilla
- Peripherally Inserted Central Catheter, Non-randomized (PICC NR): PICC non-randomized arm (observational only)
- Midline Catheter, Non-randomized (MC NR): MC non-randomized arm - observational only
Period: Overall Study
Arm/Group | Peripherally Inserted Central Catheter, Randomized (PICC R) | Midline Catheter, Randomized (MC R) | Peripherally Inserted Central Catheter, Non-randomized (PICC NR) | Midline Catheter, Non-randomized (MC NR)
Started | 4 | 4 | 6 | 21
Completed | 4 | 4 | 6 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Peripherally Inserted Central Catheter, Non-randomized (PICC NR): PICC non-randomized arm - observational only
- Midline Catheter, Non-randomized (MC NR): MC non-randomized arm -observational only
- Total: Total of all reporting groups
Arm/Group | Peripherally Inserted Central Catheter, Randomized (PICC R) | Midline Catheter, Randomized (MC R) | Peripherally Inserted Central Catheter, Non-randomized (PICC NR) | Midline Catheter, Non-randomized (MC NR) | Total
Number analyzed (Participants) | 4 | 4 | 6 | 21 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.2 [4.0 to 16.8] | 10.8 [4.5 to 16.3] | 8.4 [6.2 to 15.8] | 11.2 [7.7 to 15.0] | 9.8 [6.2 to 15.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 2 | 9 | 15
  Male | 0 | 4 | 4 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 3 | 2 | 6 | 19 | 30
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 2 | 3
  White | 3 | 3 | 6 | 17 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Severity/Location [Count of Participants; unit: Participants]
  Acute care | 4 | 4 | 6 | 11 | 25
  Critical care | 0 | 0 | 0 | 10 | 10
Primary Diagnosis [Count of Participants; unit: Participants]
  Medical | 4 | 4 | 4 | 5 | 17
  Surgical | 0 | 0 | 2 | 16 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent Eligible Patients That Agreed to Participate
Description: Percent eligible patients that agreed to participate in the randomized part of the study
Time Frame: Day of enrollment
Population: The primary outcome, a feasibility outcome, only applied to the randomized portion of the study (PICC R and MC R arms); and is the proportion of patients that agreed to participate in randomization out of all eligible patients. Therefore, the Overall Number of Participants Analyzed represents the number of participants eligible for the randomization part of the study prior to enrollment.
Measure: Number; unit: percentage of eligible patients agreed t
Groups:
- Eligible Participants: All participants eligible for the randomized portion of the study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 10
percentage of eligible patients agreed t | 80

2. Primary Outcome: Average Dwell-time
Description: Dwell-time will be measured using the time-to-device removal for all reasons (both secondary to completion of therapy and secondary to complications).
Time Frame: An average of 14 days
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Midline Catheter, Randomized (PICC R): MC Randomized arm:
  An uncoated MC with available sizes of 8 cm, 20 to 22G (Powerglide, Becton Dickinson). The catheter size was selected by an inserter based on patient size. All MCs were placed in the upper arm with the tip of the catheter ending at or below the axilla
Arm/Group | Peripherally Inserted Central Catheter, Randomized (PICC R) | Midline Catheter, Randomized (PICC R) | Peripherally Inserted Central Catheter, Non-randomized (PICC NR) | Midline Catheter, Non-randomized (MC NR)
Number analyzed (Participants) | 4 | 4 | 6 | 21
days | 11.0 [7.8 to 12.0] | 4.7 [3.3 to 5.9] | 8.5 [5.5 to 18.9] | 8.0 [6.2 to 9.1]

3. Secondary Outcome: Number of Participants Who Completed Therapy With Initial VAD
Description: percent of participants in each group that completed the therapy the VAD was requested for with original VAD
Time Frame: An average of 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Peripherally Inserted Central Catheter, Randomized (PICC R) | Midline Catheter, Randomized (MC R) | Peripherally Inserted Central Catheter, Non-randomized (PICC NR) | Midline Catheter, Non-randomized (MC NR)
Number analyzed (Participants) | 4 | 4 | 6 | 21
Participants | 4 | 1 | 6 | 15

4. Secondary Outcome: Number of Participants With at Least One Complications
Description: the rate of any complications, including suspected VTE (ultrasound obtained), suspected CLABSI (blood culture obtained), confirmed VTE (ultrasound positive for clot), confirmed CLABSI (blood culture positive), dislodgement, occlusion, phlebitis, line dysfunction, infiltration, leaking
Time Frame: An average of 14 days
Measure: Count of Participants; unit: Participants
Groups:
- PICC R: PICC Randomized arm:
  An uncoated polyurethane PICC with an external clamp was placed in the upper arm, and the available sizes were 3 to 6Fr (Bard, Becton Dickinson). The catheter type and size were selected based on IR standard protocol.
- MC R: MC Randomized arm:
  An uncoated MC with available sizes of 8 cm, 20 to 22G (Powerglide, Becton Dickinson). The catheter size was selected by an inserter based on patient size. All MCs were placed in the upper arm with the tip of the catheter ending at or below the axilla
- PICC NR: PICC non-randomized arm (observational only)
- MC NR: MC non-randomized arm - observational only
Arm/Group | PICC R | MC R | PICC NR | MC NR
Number analyzed (Participants) | 4 | 4 | 6 | 21
Participants | 2 | 3 | 3 | 8

5. Secondary Outcome: Number of Participants That Received Sedation for VAD Placement
Description: sedation completed (yes/no)
Time Frame: 1 day (day of enrollment/VAD placement)
Measure: Count of Participants; unit: Participants
Arm/Group | PICC R | MC R | PICC NR | MC NR
Number analyzed (Participants) | 4 | 4 | 6 | 21
Participants | 4 | 3 | 5 | 18

6. Secondary Outcome: Number of Participants With VAD Successfully Used for Blood Draws
Description: at least one successful blood draw (yes/no)
Time Frame: An average of 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | PICC R | MC R | PICC NR | MC NR
Number analyzed (Participants) | 4 | 4 | 6 | 21
Participants | 4 | 2 | 5 | 10

7. Secondary Outcome: Number of Participants Requiring Additional VADs to Complete Therapy
Description: any additional VADs placed to complete therapy or supplement therapy
Time Frame: An average of 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | PICC R | MC R | PICC NR | MC NR
Number analyzed (Participants) | 4 | 4 | 6 | 21
Participants | 0 | 3 | 1 | 4

ADVERSE EVENTS:
Time Frame: Up to 1 month while catheter in place
Description: We report catheter-related confirmed VTE (ultrasound results positive for clot at catheter site), confirmed CLABSI (defined using the National Healthcare Safety Network surveillance definition)
Arm/Group | PICC R | MC R | PICC NR | MC NR
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/6 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/6 | 0/21
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 0/6 | 5/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PICC R (N=4) | MC R (N=4) | PICC NR (N=6) | MC NR (N=21)
Occlusion (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Infiltration (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Dislodgement (Product Issues) | 0 | 0 | 0 | 2
Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT05346406/Prot_SAP_000.pdf